CLINICAL TRIAL: NCT06460701
Title: Effects of Modified Constraint Induced Movement Therapy With and Without Kinesiotaping for Children With Erb's Palsy
Brief Title: Effects of m-CIMT With and Without Kinesiotaping for Children With Erb's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/07104
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Erb Palsy
Keywords: Erb's Palsy ,; mCIMT; Kinesiotaping; OBPI .
MeSH Terms: conditions — Brachial Plexus Neuropathies

STUDY DESIGN:
Intervention Model Description: it will be a randomized controlled trial in which non probability convenient sampling will be used. Two groups of 2-4 age will be formed in which participants will be randomly divided. Group A will receive m-CIMT along with kinesio taping while Group B will receive only m-CIMT.
Who Masked: Participant
Masking Description: participants will get separate treatment protocols and possible efforts will be put to mask both groups about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active comparator: modified constraint induced movement therapy without Kinesiotaping. (Active Comparator): in this group m-CIMT will be applied without kinesiotaping.
  Interventions: Other: m-CIMT without Kinesio taping
- Experimental: modified constraint induced movement therapy along with kinesio taping. (Experimental): in this group m-CIMT will be applied along with kinesiotaping.
  Interventions: Other: m-CIMT along with kinesiotaping

INTERVENTIONS:
Other: m-CIMT without Kinesio taping — Baseline treatment m-CIMT will be applied includeing ROM with a sling, e.g shoulder flexion, extension, abduction, and rotation. The elbow's flexion and extension, Forearm supination is the extension of the wrist and fingers. Functional Training Using a tiny toy ball, practice tossing and catching it from various angles. Play with modeling clay, constructing towers of the toy bricks using LEGOs,Using crayons, ripping a piece of paper towel,Grasping biscuits, Using a spoon, utilizing a glass to drink, comb hair, brush teeth,Using a bubble blower,With a toy in hand, putting cap, putting lotion.stretching to shoulder's extensors, adductor, and internal rotators ,wrist and elbow flexors. strengthening exercises e.g a ball above head position in various directions,Using paper adhered to the window or wall at varying heights for drawing. The session will go for one hour.
  Arms: Active comparator: modified constraint induced movement therapy without Kinesiotaping.
Other: m-CIMT along with kinesiotaping — Modified constraint-induced movement therapy along with kinesiotaping will be applied. m-CIMT protocol is baseline treatment and it is is same as in the other group.
  This group also participated additionally in a kinesio taping program, which utilize KT with the goal of enhancing middle and lower trapezius function to increase stability in the scapula on the afflicted side. During the application of the tape, the shoulders were kept in a low and backward posture, and the scapular alignment was manually maintained. KT was administered at the acromion and positioned medially at the spinous processes (T2-T3 for the middle trapezius and T12 for the lower trapezius). For eight weeks in a row, there will be three sessions every week
  Arms: Experimental: modified constraint induced movement therapy along with kinesio taping.

SUMMARY:
The upper brachial plexus, a network of nerves in the neck and shoulder, is affected by Erb's palsy, often referred to as Erb-Duchenne palsy. This syndrome usually arises after labor, particularly if the baby's head and neck are pulled or stretched excessively during delivery. Erb's palsy can cause the hand and arm on the afflicted side of the body to become paralyzed or feeble. Erb's palsy symptoms can include: restricted range of motion in the injured arm. weakened hand and arm in the afflicted area, loss of feeling in the hand or arm. The effected arm is in "waiter's tip" position in which the elbow is bent and the wrist is flexed. The purpose of this research is to evaluate the effectiveness of modified constraint-induced movement therapy in children with erb's palsy, both with and without kinesiotaping.

Convenient sampling will be the method of sampling, and the study design will be randomized control trial. There will be two groups created with n = 40 subjects each. Twenty participants will be divided into two groups: twenty for each group will receive modified constraint-induced movement therapy plus kinesiotaping, while twenty for the other group will receive modified constraint-induced movement therapy alone. The youngsters will be evaluated using the Active Movement Scale.Both at the program's baseline and after the intervention is over, data will be gathered. The course of treatment will run for eight weeks straight, meeting three times a week for an hour each time. Based on inclusion criteria, subjects from Ayesha Amir Memorial Hospital and Children Hospital Faisalabad will be chosen. Data analysis will be done using SPSS 25.00.

DETAILED DESCRIPTION:
Group A will be applied modified constraint induced movement therapy , session will last for one hour including following exercises such as ROM with the sling. Flexion, extension, abduction, and rotation of the shoulder. Flexion and extension of the elbow, Supination of forearm-Extension of wrist and finger. Stretching exercises for internal rotators , adductors ,extensors of shoulder. This will reduce the tightness and enhance the range of movement. Strengthening exercises also be applied to this group by throwing a ball in different directions above head position ,by drawing on paper stuck on the wall or window at different heights, by supinating bottles weighing <500g as tolerated by the child by thera band exercises above, across, and below the chest. Repetitive movement such as supinating the light bottles. Functional activities including some playful movement will be done by this group in which children are involved in different activities e.g playing with toys, blocks and such objects. Additionally, this group will engaged in a kinesiotaping program which aims to obtain more stability to the scapula on the affected side through facilitating middle and lower trapezius function. The shoulders will be kept in downward and back- ward position, while the alignment of scapulae should be manually maintained during the tape application. KT will set medially at the spinous processes (T2-T3 for middle trapezius and T12 for lower trapezius) and will be applied toward the acromion.

Group B will undergo same intervention such as group A alongwith m-CIMT but without the application of kinesiotaping.

There will be three sessions per week for the eight consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age of 2 years to 4 years.
* Children with Erb's palsy.
* Healthy BMI, ability to understand the command
* No previous mCIMT and kinesiotaping intervention was given

Exclusion Criteria:

* Children with visual deficits,
* Children with seizures or epilepsy,
* systemic disease or infectious disease,
* children with permanent arm deformities

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-06-16 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Active Movement Scale | 8 weeks
  Active Movement Scale (AMS) is a unique assessment instrument that may be applied to children and newborns at any stage of development.. Tests are conducted for flexion, external rotation, internal rotation, abduction, and adduction of the shoulder, flexion and extension of the elbow, pronation and supination of the forearm, and flexion and extension of the wrist, finger, and thumb. AMS is measured on an 8-point scale (0 for no discernible contraction and 7 for full motion). For correct scoring, it is advised that the estimated passive range of motion (PROM) be confirmed using goniometry. Using kappa statistics, the scores were examined for reliability and chance agreement was managed. The 15 tested movements' overall kappa analysis revealed a moderate degree of score agreement (kappa = 0.51). Eight of the fifteen movements examined fell into the highest strength of agreement group (kappa(quad) = 0.81-1.00), according to quadratic-weighted kappa (kappa(quad)) statistics. Two movements
Goniometer | 8 weeks
  A goniometer is a specialized tool used in physical therapy that measures and evaluates the range of motion (ROM) of joints in the human body. Physical therapists and other medical professionals use it as a vital tool for diagnosing, treating, and keeping track of a variety of musculoskeletal injuries, diseases, and rehabilitation processes. The findings showed good intra-rater reliability between sessions (ICC2,1 = 0.83 to 0.98), across sessions (ICC2,2 = 0.79 to 0.97), and high inter-rater reliability between sessions (ICC2,2 = 0.79 to 0.92).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Zaheer, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuran B, Azrak SD, Dogu B, Yilmaz F, Sirzai H, Oncu J, Terlemez R, Ayyildiz A. The Effect of the Modified Constraint-Induced Movement Therapy on the Upper Extremity Functions of Obstetric Brachial Plexus Palsy Patients. Sisli Etfal Hastan Tip Bul. 2022 Dec 19;56(4):525-535. doi: 10.14744/SEMB.2022.32956. eCollection 2022. PMID 36660395